CLINICAL TRIAL: NCT00169364
Title: Comparison of Clinical, Molecular and Metabolic Characteristics of PD Patients With and Without Parkin Mutation
Brief Title: Clinical, Molecular and Metabolic Characteristics of Parkinson's Disease (PD) Patients With Parkin Mutation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Collaborators: University Hospital, Tours (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P011104
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2007-08-29 (Estimated); Status verified 2005-09

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; parkin mutation; Juvenile parkinson's disease; positron emission tomography
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders | interventions — Positron-Emission Tomography

INTERVENTIONS:
Device: positron emission tomography

SUMMARY:
Parkinson's disease is a frequent neurodegenerative disorder. Genetic forms of the disease have been recently identified. The monogenic form due to parkin mutation is responsible for many familial cases and sporadic forms. However, the relationship between the mutation and the genotype of patients is not fully established. The aim of this study is to compare clinical, metabolic and neuropsychological characteristics obtained in patients with parkin mutation with those of patients without parkin mutation.

ELIGIBILITY:
Inclusion Criteria:

* Juvenile Parkinson's disease (< 45 years)
* Parkin mutation
* Normal brain magnetic resonance imaging (MRI)

Exclusion Criteria:

* Contraindication to brain MRI
* Women without effective contraception

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2002-05

PRIMARY OUTCOMES:
Parkin mutation
Motor disability
Neuropsychological evaluation
Psychiatric evaluation

SECONDARY OUTCOMES:
Positron emission tomography

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Brice, MD, PhD, Study Director — Groupe Hospitalier Pitié-Salpêtrière
Locations (1):
- Centre d'Investigation Clinique-Hôpital Pitié-Salpetriere, Paris, France